CLINICAL TRIAL: NCT01455103
Title: A Phase I Study of the Biologic Effects of BMS-936559 Treatment in Subjects With Unresectable Stage III or IV Melanoma
Brief Title: Phase 1 Biomarker Study of Anti-PDL-1 in Advanced Melanoma
Acronym: PD-L1
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CA210-002
Record Dates: First submitted 2011-10-18; First posted 2011-10-19 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-10

CONDITIONS: Stage III or IV Melanoma
MeSH Terms: interventions — BMS-936559

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: BMS-936559 (1mg/kg) (Experimental)
  Interventions: Biological: BMS-936559 (Anti-PD-L1)
- Arm 2: BMS-936559 (3mg/kg) (Experimental)
  Interventions: Biological: BMS-936559 (Anti-PD-L1)
- Arm 3: BMS-936559 (10mg/kg) (Experimental)
  Interventions: Biological: BMS-936559 (Anti-PD-L1)

INTERVENTIONS:
Biological: BMS-936559 (Anti-PD-L1) — Solution, Intravenous infusion, 1 mg/kg, Every 2 weeks, Up to 2 years, depending on response
  Other Names: MDX1105
  Arms: Arm 1: BMS-936559 (1mg/kg)
Biological: BMS-936559 (Anti-PD-L1) — Solution, Intravenous infusion, 3 mg/kg, Every 2 weeks, Up to 2 years, depending on response
  Other Names: MDX1105
  Arms: Arm 2: BMS-936559 (3mg/kg)
Biological: BMS-936559 (Anti-PD-L1) — Solution, Intravenous infusion, 10 mg/kg, Every 2 weeks, Up to 2 years, depending on response
  Other Names: MDX1105
  Arms: Arm 3: BMS-936559 (10mg/kg)

SUMMARY:
The purpose of this study is to evaluate pharmacodynamic changes of BMS-936559 treatment on the biomarkers measured in the peripheral blood and tumor tissues of subjects with unresectable Stage III or IV Melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) status = 0 to 1
* Subjects with unresectable Stage III or IV Melanoma who are either refractory or intolerant to, or have refused standard therapy for treatment of metastatic Melanoma
* Subject must have histologic or cytologic confirmation of advanced Melanoma
* Subjects must have at least one measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Subjects must have at least 1 tumor site that can be biopsied at acceptable clinical risk and must consent to pre- and post-treatment biopsies

Exclusion Criteria:

* Active or progressing brain metastases
* Other concomitant malignancies (with some exceptions per protocol)
* Active or history of autoimmune disease
* Positive test for human immunodeficiency virus (HIV) 1&2 or known acquired immunodeficiency syndrome (AIDS)
* History of any hepatitis
* Prior therapy with any antibody/drug that targets the T cell coregulatory proteins, including but not limited to, anti Programmed cell death 1 (PD-1), anti Programmed cell death ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40 or anti Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Evidence of immunomodulatory effects of BMS-936559 as measured by changes from baseline in biomarkers assessed 1) peripheral blood assays including flow cytometry and soluble factors and 2) tumor based assays including immunohistochemistry | Baseline and within the first 24 weeks of study participation

SECONDARY OUTCOMES:
Safety and tolerability of BMS-936559 as measured by the incidence of adverse events (AEs), serious AEs, laboratory test abnormalities, and changes in vital signs | Every 2 weeks until 70 days after last treatment
Antitumor Activity of BMS-936559 as measured by the objective response rate, disease control rate, duration of response, and progression free survival | Every 6 weeks for 1 year, every 12 weeks thereafter until confirmed disease progression
Immunogenicity of BMS-936559 as measured by the frequency of subjects with an increase in anti-drug antibody levels from baseline | Baseline, Week 6, Week 12, and then every 12 weeks until follow-up
Pharmacodynamic activity of BMS-936559 as measured by changes from baseline of the tetramer assay in HLA-A*0210 positive subject only | Predose (screening) and Cycle 3 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb